CLINICAL TRIAL: NCT01059409
Title: The Clinical and Medico-economical Evaluation of Meniscal Allografts in the Sequelae of Total or Sub-total Meniscectomy.
Brief Title: Study of Meniscal Allografts
Acronym: ERAM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient number of patients included compared to the expected duration of inclusion.
  sponsor's decision
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P070309 / IC0705
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-03

CONDITIONS: Meniscectomy Sequelae
Keywords: Meniscal Allografts; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meniscal Allograft (Experimental)
  Interventions: Procedure: Meniscal Allograft

INTERVENTIONS:
Procedure: Meniscal Allograft — Meniscal Allograft

SUMMARY:
Total or subtotal meniscectomies in young patients are currently responsible of pain and limitation of activities. There isn't any other treatment than meniscal replacement. But there is no randomized clinical trial on meniscal allograft to validate the efficiency of this treatment.

DETAILED DESCRIPTION:
Meniscal allograft is done through United States and Europe since the last fifteen years. Operative technique has regularly improved, especially because of new arthroscopic devices. The meniscal allografts to be used are taken from dead donors and then frozen according to all the reglementary aspects of tissue bank.

The graft has to be ordered as soon as the patient is randomized ; the sizing of the graft ordered is important depending on the gender size and height of the patient and on the measures of the tibial plateau on X Rays.

The arthroscopic procedure is done under general or loco-regional anesthesia. The graft has to be prepared with bone blocks attached to the anterior and posterior horn of the meniscal graft. These bone blocks will be fixed through bone tunnels and the meniscus itself will be sutured on the peripheral meniscus synovial rim.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 on
* Previous total or subtotal meniscectomy
* Medical insurance
* Female patients have to be under contraceptive treatment
* Sign consent form

Exclusion Criteria:

* Age < 18 years
* Pregnant or breast-feeding woman
* Need of a simultaneous frontal osteotomy
* Inflammatory disease
* Septic background
* Psychiatric background
* Understanding difficulties or problems for follow-up
* No consent
* No medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
"Function" Subscale in the Koos Scale (area under the curve) | 2 years follow up
  Koos Scale

SECONDARY OUTCOMES:
Clinical criteria: pain, quality of life, professional activity | At 2 years follow-up
  Pain, quality of life, professional activity
Post operative and late complications | At 2 years follow-up
  Post operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Patricia THOREUX, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - POTEL Jean-François, Clinique Medipole Garonne, Toulouse
  - Hôpital Avicenne - Service de Chirurgie orthopédique, Bobigny, Île-de-France Region